CLINICAL TRIAL: NCT00837083
Title: Open-Label Non-Interventional Evaluation of Efficacy of Crestor® (Rosuvastatin) in Reduction of LDL-Cholesterol and Cardiovascular Risk Parameters in Patients With Hypercholesterolaemia
Brief Title: Evaluation of Crestor® (Rosuvastatin) in Daily Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Meta Jeras; Regulatory and Medical Affairs Manager, AstraZeneca
Other Study IDs: NIS-CSI-CRE-2006/1; NIS-CRE 01/06
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; cholesterol; LDL-cholesterol; rosuvastatin; Crestor
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This open label, non-interventional study is to show the efficacy of Crestor (rosuvastatin) in reduction of LDL-cholesterol and cardiovascular risk parameters in patients with hypercholesterolemia. Effectiveness is to be evaluated using the difference in LDL cholesterol level between the first and the second visit after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* a patient with hypercholesterolemia who has been prescribed Crestoraccording to physician's judgement, irrespective of the inclusion in the study.
* no treatment with any statin in the last 3 months

Exclusion Criteria:

* hypersensitivity to rosuvastatin or any other ingredient of Crestor
* active liver disease, severe renal insufficiency
* myopathy or predisposing risk factors for myopathy/ rhabdomyolysis
* woman of child-bearing potential and not using appropriate contraceptive measures, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients (outpatient or hospitalised) in whom Crestor is indicated according to the current Summary of product characteristics (SPC)
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol reduction | 12 weeks

SECONDARY OUTCOMES:
achievement of target levels of total cholesterol and LDL-cholesterol | 12 weeks
patient compliance | 12 weeks
change in coronary risk | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matija Cevc, MD, Principal Investigator — University Medical Centre Ljubljana